CLINICAL TRIAL: NCT06158958
Title: A Phase 1 First-in-Human, Open-Label Study Evaluating the Safety, Pharmacokinetics, and Efficacy of ABBV-303, as Monotherapy and in Combination With Budigalimab (ABBV-181), in Adult Subjects With Advanced Solid Tumors
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Efficacy of Intravenous (IV) ABBV-303, as Monotherapy and in Combination With IV Infused Budigalimab (ABBV-181), in Adults With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-122; 2023-504714-30 (Other: EU CT)
Record Dates: First submitted 2023-11-29; First posted 2023-12-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Non-Small Cell Lung Cancer; NSCLC; Renal Cell Carcinoma; RCC; Head and Neck Squamous Cell Carcinoma; HNSCC; ABBV-303; ABBV-181; Budigalimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- ABBV-303 Dose Escalation: Part 1A Monotherapy (Experimental): Participants with (R)/refractory (R) solid tumors will receive ABBV-303 in escalating doses as a monotherapy until the maximum tolerable dose (MTD) is determined as part of the 3 year study duration.
  Interventions: Drug: ABBV-303
- ABBV-303 Dose Expansion: Part 2A Monotherapy (Experimental): Participants with R/R NSCLC will receive ABBV-303 at the recommended phase 1 expansion dose (RP1ED) as a monotherapy as part of the 3 year study duration.
  Interventions: Drug: ABBV-303
- ABBV-303 Dose Expansion: Part 3A Monotherapy (Experimental): Participants with R/R RCC will receive ABBV-303 at the RP1ED as a monotherapy as part of the 3 year study duration.
  Interventions: Drug: ABBV-303
- ABBV-303 Dose Expansion: Part 4A Monotherapy (Experimental): Participants with R/R HNSCC will receive ABBV-303 at the RP1ED as a monotherapy as part of the 3 year study duration.
  Interventions: Drug: ABBV-303
- ABBV-303 Dose Expansion: Part 5A Monotherapy (Experimental): Tissue agnostic with R/R participants with MET amplification by any commercially available test will receive ABBV-303 at the RP1ED as a monotherapy as part of the 3 year study duration.
  Interventions: Drug: ABBV-303
- ABBV-303 Dose Escalation: Part 1B Combination (Experimental): Participants with R/R solid tumors will receive ABBV-303 in combination with budigalimab at or below the MTD as part of the 3 year study duration.
  Interventions: Drug: ABBV-303; Drug: Budigalimab
- ABBV-303 Dose Expansion: Part 2B Combination (Experimental): Participants with R/R NSCLC will receive ABBV-303 at or below the MTD in combination with budigalimab as part of the 3 year study duration.
  Interventions: Drug: ABBV-303; Drug: Budigalimab

INTERVENTIONS:
Drug: ABBV-303 — Intravenous (IV) Infusion
Drug: Budigalimab — IV Infusion
  Other Names: ABBV-181
  Arms: ABBV-303 Dose Escalation: Part 1B Combination; ABBV-303 Dose Expansion: Part 2B Combination

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess safety, tolerability, pharmacokinetics and preliminary efficacy of ABBV-303 as a monotherapy and in combination with budigalimab, (ABBV-181).

ABBV-303 is an investigational drug being developed for the treatment of solid tumors. There are multiple treatment arms in this study. Participants will either receive ABBV-303 as a single agent or in combination with budigalimab (another investigational drug) at different doses. Approximately 181 adult participants will be enrolled in the study across sites worldwide.

In Part A, ABBV-303 will be intravenously (IV) infused in escalating doses as a monotherapy in participants with relapsed (R)/refractory (R) solid tumors, R/R non-small cell lung cancer (NSCLC), R/R renal cell carcinoma (RCC), R/R head and neck squamous cell carcinoma (HNSCC), or R/R tissue agnostic participants with mesenchymal epithelial transition. In Part B, ABBV-303 in combination with budigalimab will be IV infused in participants with R/R solid tumors or NSCLC. The estimated duration of the study is up to 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Laboratory values meeting the protocol's criteria within the screening period (-28 days) prior to the first dose of study drug.
* Participants with a diagnosis of a malignant solid tumor by histology (World Health Organization [WHO] criteria).
* Participants with measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

Exclusion Criteria:

* Unresolved Grade > 1 adverse events (AEs) from prior anti-cancer therapy except for alopecia.
* Active systemic or uncontrolled local bacterial, fungal, or viral infection requiring antimicrobial therapy.
* History of hypersensitivity to the active ingredients or any excipients of ABBV-303 and budigalimab (ABBV-181).
* Body weight < 35 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AE) | Up to 3 Years
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 3 Years
  ORR defined as percentage of participants with confirmed best overall response of Confirmed complete response (CR) and partial response (PR) per investigator review according to RECIST version 1.1.
Duration of Response (DOR) for Participants with Confirmed CR/PR per RECIST v1.1 | Up to 3 Years
  DOR is defined for participants achieving a confirmed CR+PR as the time from the initial response of CR+PR per investigator review according to RECIST 1.1 criteria to disease progression or death of any cause, whichever occurs earlier.
Progression-free survival (PFS) | Up to 3 Years
  PFS is defined as time from first study treatment to a documented disease progression according to RECIST version 1.1, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall survival (OS) | Up to 3 Years
  OS is defined as time from first study treatment to death due to any cause.
ORR per Immune-Mediated Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 3 Years
  ORR defined as percentage of participants with confirmed best overall response of Confirmed complete response (CR) and partial response (PR) per investigator review according to iRECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- United States (11):
  - City of Hope /ID# 254303, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 266792, Irvine, California
  - University of Southern California /ID# 254356, Los Angeles, California
  - START Midwest /ID# 256945, Grand Rapids, Michigan
  - Washington University-School of Medicine /ID# 262943, St Louis, Missouri
  - NYU Langone - Laura and Isaac Perlmutter Cancer Center /ID# 256943, New York, New York
  - Carolina BioOncology Institute /ID# 254305, Huntersville, North Carolina
  - The Ohio State University - The James /ID# 260475, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center /ID# 254308, Houston, Texas
  - NEXT Oncology /ID# 257395, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics /ID# 256944, San Antonio, Texas
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 259408, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 254608, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 254606, Jerusalem
- Japan (4):
  - National Cancer Center Hospital East /ID# 261712, Kashiwa-shi, Chiba
  - Shizuoka Cancer Center /ID# 261714, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 254359, Chuo-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 254361, Wakayama, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-122